CLINICAL TRIAL: NCT06276777
Title: The Effect of Using Desensitizers Containing S-PRG Versus Sodium Fluoride With Functionalized Tri-Calcium Phosphate In Treatment Of Dentin Hypersensitivity In Adult Patients Over 6 Months: A Randomized Clinical Trial
Brief Title: The Effect of Using Desensitizers Containing S-PRG In Treatment Of Dentin Hypersensitivity Over 6 Months: A Randomized Clinical Trial
Acronym: S-PRG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eman Omar Elfarouk (Other)
Responsible Party: Sponsor-Investigator, Eman Omar Elfarouk, masters degree student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPRG Dentin Hypersensitivity
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Dentin Hypersensitivity
Keywords: S-PRG
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and both assessors will be blind to the type of material used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varnish contains S-PRG (PRG Barrier Coat from Shofu) (Experimental): Treatment of dentin hypersensitivity by application of tooth varnish containing S-PRG.
  Interventions: Procedure: Tooth varnish (PRG Barrier Coat from Shofu)
- Varnish contains sodium fluoride and functionalized tri-calcium phosphate(Clinpro white varnish 3M) (Active Comparator): Treatment of dentin hypersensitivity by application of tooth varnish containing sodium fluoride with functionalized tri-calcium phosphate.
  Interventions: Procedure: Tooth varnish (Clinpro white varnish 3M)

INTERVENTIONS:
Procedure: Tooth varnish (PRG Barrier Coat from Shofu) — Treatment of cervical dentin hypersensitivity with tooth desensitizers.
  Arms: Varnish contains S-PRG (PRG Barrier Coat from Shofu)
Procedure: Tooth varnish (Clinpro white varnish 3M) — Treatment of cervical dentin hypersensitivity with tooth desensitizers.
  Arms: Varnish contains sodium fluoride and functionalized tri-calcium phosphate(Clinpro white varnish 3M)

SUMMARY:
The goal of this clinical trial is to compare the effect of desensitizer containing S-PRG have similar effect as sodium fluoride with functionalized tri-calcium phosphate containing desensitizer in relieving dentinal hypersensitivity in adult patients for six months follow-up. patients will be asked to report pain degree on the visual analogue scale (VAS) along the follow up periods on both groups.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene.
* Cooperative patients who show interest to participate in the study and welling to sign the informed consent.
* Healthy patients with no history of previous systematic diseases that can affect their oral health.
* Normal and healthy gingival tissue.
* Teeth that have no cavitation or restorations.
* Patients with at least 20 natural permanent teeth and at least two teeth with a VAS score from 4 to 10.
* Anterior teeth.

Exclusion Criteria:

* Allergic to the ingredients used in the study.
* Gastrointestinal disorders (They have repeated vomiting attacks).
* Medically compromised (They cannot tolerate the procedures).
* Taking desensitizing treatment in the last 6 months (It affects the outcome).
* Taking anti-inflammatory drugs (It affects the hypersensitivity perception).
* Pregnant females (They complain from nausea and repeated vomiting attacks)
* Smokers (Smoking will affect the oral hygiene and periodontal health).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Dentin hypersensitivity reduction | assessment will be done immediately after the treatment then after 1 week, 4 weeks, 3 months and 6 months.
  The participants will point out the degree of sensitivity on the VAS scale (0-10) chart.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omar, bachelor, Principal Investigator — Cairo University faculty of oral and dental medicine
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No